CLINICAL TRIAL: NCT01677286
Title: A Phase II Study of Doxycycline in Patients With Amyloidosis
Brief Title: Safety and Effect of Doxycycline in Patients With Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, John L. Berk, Assistant Director, Amyloidosis Center, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31546
Record Dates: First submitted 2012-08-21; First posted 2012-09-03 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Amyloidosis
Keywords: AL Amyloidosis; Primary Amyloidosis; Hereditary Amyloidosis; Familial Amyloidosis; SSA Amyloidosis; Senile Systemic Amyloidosis; AA Amyloidosis; Secondary Amyloidosis; Localized Amyloidosis; Systemic Amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis; Amyloidosis, Familial; AA amyloidosis | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- doxycycline 100 mg po bid x 12 months (Experimental): Open-label doxycycline 100 mg twice daily by mouth will be administered to subjects for 12 months.
  Interventions: Drug: Doxycycline 100 mg po bid x 12 months

INTERVENTIONS:
Drug: Doxycycline 100 mg po bid x 12 months — 100mg by mouth twice daily for 1 year.
  Other Names: CAS: 564-25-0; ATC code: J01AA02 A01AB22; PubChem: CID 11256

SUMMARY:
The tetracycline antibiotic doxycycline disrupts A beta amyloid fibrils (AB) in Alzheimer's disease, transthyretin (ATTR) amyloid fibrils in familial amyloidotic polyneuropathy, and immunoglobulin light chain (AL) amyloid fibrils in transgenic mouse models of disease. If untreated, amyloid deposits impair organ function, affecting the morbidity and mortality of patients.

This single-center, twelve-month, open-label, prospective, pilot phase II study aims to determine whether doxycycline reduces amyloid deposits and improves organ function in patients with systemic or localized amyloidosis.

The investigators plan to enroll patients with measurable amyloid disease according to internationally-accepted diagnostic criteria. Patients must have stable organ function at enrollment. Eligible subjects not receiving active treatments for amyloidosis affecting their kidneys, heart, aerodigestive tracts, peripheral or autonomic nervous system(s), lungs, eyes, skin, bladder, or breasts will undergo evaluations at baseline, 6 months, and 12 months - or more frequently as clinically indicated.

Over 45 years experience indicates doxycycline is a safe, well tolerated antibiotic. The investigators will use standard grading systems to assess doxycycline response following twelve months of treatment.

DETAILED DESCRIPTION:
In transgenic animal models of disease, the tetracycline antibiotic doxycycline disrupts A beta amyloid fibrils (AB) in Alzheimer's disease, transthyretin (ATTR) amyloid fibrils in familial amyloidotic polyneuropathy, and immunoglobulin light chain (AL) amyloid fibrils.

The aim of this single-center, 12-month open label, prospective phase II study was to determine a) the safety and tolerability of prolonged full dose doxycycline in patients with amyloidosis, and b) the effect of doxycycline treatment on amyloid-induced organ dysfunction.

We enrolled 25 patients with measurable organ dysfunction caused by amyloid deposition who were not receiving active treatment to control their amyloid production. All 25 subjects received doxycycline 100 mg by both twice daily for up to 12 months depending on their tolerance of the antibiotic. The primary endpoint, defined by the organ most affected by amyloid, was measured at baseline, 6 and 12 months along with safety laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Biopsy-proven amyloidosis
* Biochemical or clinical evidence of amyloid induced end-organ dysfunction

Exclusion Criteria:

* Concurrent use of other tetracyclines
* Ongoing active treatment for amyloidosis
* Pregnancy or unwillingness to use contraception by women of childbearing age
* Doxycycline drug allergy/hypersensitivity
* ECOG performance status > 3
* NYHA class > 3
* Renal insufficiency (estimated creatinine clearance < 25 ml/min)
* Transaminitis (AST or ALT > 5 times upper limit of normal)
* Diabetes mellitus or hemoglobin A1C > 6.2%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Berk, M.D., Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Primary manuscript reporting outcomes is in preparation. Once completed, we will consider IPD sharing plan.

REFERENCES:
- [Background] Cardoso I, Merlini G, Saraiva MJ. 4'-iodo-4'-deoxydoxorubicin and tetracyclines disrupt transthyretin amyloid fibrils in vitro producing noncytotoxic species: screening for TTR fibril disrupters. FASEB J. 2003 May;17(8):803-9. doi: 10.1096/fj.02-0764com. PMID 12724338
- [Background] Cardoso I, Saraiva MJ. Doxycycline disrupts transthyretin amyloid: evidence from studies in a FAP transgenic mice model. FASEB J. 2006 Feb;20(2):234-9. doi: 10.1096/fj.05-4509com. PMID 16449795
- [Background] Forloni G, Colombo L, Girola L, Tagliavini F, Salmona M. Anti-amyloidogenic activity of tetracyclines: studies in vitro. FEBS Lett. 2001 Jan 5;487(3):404-7. doi: 10.1016/s0014-5793(00)02380-2. PMID 11163366
- [Background] Ward JE, Ren R, Toraldo G, Soohoo P, Guan J, O'Hara C, Jasuja R, Trinkaus-Randall V, Liao R, Connors LH, Seldin DC. Doxycycline reduces fibril formation in a transgenic mouse model of AL amyloidosis. Blood. 2011 Dec 15;118(25):6610-7. doi: 10.1182/blood-2011-04-351643. Epub 2011 Oct 12. PMID 21998211
- [Background] Obici L, Cortese A, Lozza A, Lucchetti J, Gobbi M, Palladini G, Perlini S, Saraiva MJ, Merlini G. Doxycycline plus tauroursodeoxycholic acid for transthyretin amyloidosis: a phase II study. Amyloid. 2012 Jun;19 Suppl 1:34-6. doi: 10.3109/13506129.2012.678508. Epub 2012 May 2. PMID 22551192
- [Background] Giorgetti S, Raimondi S, Pagano K, Relini A, Bucciantini M, Corazza A, Fogolari F, Codutti L, Salmona M, Mangione P, Colombo L, De Luigi A, Porcari R, Gliozzi A, Stefani M, Esposito G, Bellotti V, Stoppini M. Effect of tetracyclines on the dynamics of formation and destructuration of beta2-microglobulin amyloid fibrils. J Biol Chem. 2011 Jan 21;286(3):2121-31. doi: 10.1074/jbc.M110.178376. Epub 2010 Nov 10. PMID 21068391
- [Background] Cardoso I, Martins D, Ribeiro T, Merlini G, Saraiva MJ. Synergy of combined doxycycline/TUDCA treatment in lowering Transthyretin deposition and associated biomarkers: studies in FAP mouse models. J Transl Med. 2010 Jul 30;8:74. doi: 10.1186/1479-5876-8-74. PMID 20673327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred to an amyloidosis center and no longer requiring active treatment to control progressive disease were recruited to the study.
Period: Overall Study
Arm/Group | Doxycycline 100 mg po Bid x 12 Months
Started | 25
Completed | 14
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Doxycycline 100 mg po Bid x 12 Months
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: Years] | 65 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24
  Multiple | 1
  Not hispanic or latino | 24
  Unknown/not reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Brain Natriuretic Peptide (BNP) [Mean (Standard Deviation); unit: pg/mL] — Study participants with predominant cardiac amyloid involvement. Population: Patients with predominant amyloid cardiomyopathy constituted the "cardiac group" (n=12). Serial cardiac biomarkers (BNP, Troponin I) determinations were used to assess the effect of doxycycline on cardiac amyloid disease progression.
  pg/mL
    number analyzed (Participants) | 12
    (all) | 385 (294)
Troponin I [Mean (Standard Deviation); unit: ng/mL] — Study participants with predominant cardiac amyloid involvement. Population: Patients with predominant amyloid cardiomyopathy constituted the "cardiac group" (n=12). Serial cardiac biomarkers (BNP, Troponin I) determinations were used to assess the effect of doxycycline on cardiac amyloid disease progression.
  ng/mL
    number analyzed (Participants) | 12
    (all) | 0.11 (0.07)
Creatinine Clearance (mL/min) [Mean (Standard Deviation); unit: mL/min] — Study participants with predominant renal amyloid involvement. Population: Patients with predominant amyloid nephropathy constituted the "renal group" (n=10). Serial creatinine clearance and proteinuria were used to assess the effect of doxycycline on renal amyloid disease progression.
  mL/min
    number analyzed (Participants) | 10
    (all) | 83.3 (36.5)
Proteinuria (g/day) [Mean (Standard Deviation); unit: g/day] — Study participants with predominant renal amyloid involvement. Population: Patients with predominant amyloid nephropathy constituted the "renal group" (n=10). Serial creatinine clearance and proteinuria were used to assess the effect of doxycycline on renal amyloid disease progression.
  g/day
    number analyzed (Participants) | 10
    (all) | 5.99 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Amyloid Cardiomyopathy: BNP
Description: Cardiac biomarkers (BNP, Troponin I) were assessed at baseline, 6 and 12 months, with change at end of study reported
Time Frame: 12 months
Population: Analysis is limited to the patients with predominant amyloid heart involvement at enrollment. Mixed models analyses of change from baseline levels of cardiac biomarkers (BNP, Troponin I) were performed to include all collected data.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Cardiomyopathy: Patients with predominant amyloid involvement of the heart.
Arm/Group | Cardiomyopathy
Number analyzed (Participants) | 12
pg/mL | 883 (703)
Statistical Analysis 1: Comparison: Cardiomyopathy; BNP pg/mL, baseline versus end study values; Test type: Other — P-values and confidence intervals are not adjusted for multiple testing; p = 0.035, Mixed Models Analysis; degrees of freedom = 12; Mean outcome change = 171, 95% CI 2-sided [14.1 to 328]

2. Primary Outcome: Amyloid Cardiomyopathy: Troponin I
Description: Cardiac biomarkers (BNP, Troponin I) were assessed at baseline, 6 and 12 months, with change at change at end of study reported
Time Frame: 12 months
Population: Patients with predominant amyloid involvement of the heart.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardiomyopathy
Number analyzed (Participants) | 12
ng/mL | 0.15 (0.07)
Statistical Analysis 1: Comparison: Cardiomyopathy; Troponin I ng/mL, baseline versus end study levels; Test type: Other — P-values and confidence intervals are not adjusted for multiple testing; p = 0.340, Mixed Models Analysis; degrees of freedom = 12; Mean outcome change = 0.0072, 95% CI 2-sided [-0.009 to 0.0234]

3. Primary Outcome: Amyloid Nephropathy: Creatinine Clearance
Description: Creatinine clearance (ml/min) and proteinuria (g/day) were assessed at baseline, 6 and 12 months, with change at change at end of study reported
Time Frame: 12 months
Population: Analysis is limited to the patients with predominant amyloid kidney involvement at enrollment. Mixed models analyses of change from baseline levels of creatinine clearance (ml/min) and proteinuria (g/day) were performed to include all collected data.
Measure: Mean (Standard Deviation); unit: ml/min
Groups:
- Amyloid Nephropathy: Patients with predominant amyloid kidney involvement at enrollment.
Arm/Group | Amyloid Nephropathy
Number analyzed (Participants) | 10
ml/min | 82.4 (48.0)
Statistical Analysis 1: Comparison: Amyloid Nephropathy; Creatinine clearance, baseline versus end study levels; Test type: Other — P-values and confidence intervals are not adjusted for multiple testing; p = 0.017, Mixed Models Analysis; degrees of freedom = 10; Change in outcome measure = -7.39, 95% CI 2-sided [-13.12 to -1.67]

4. Primary Outcome: Amyloid Nephropathy: Proteinuria
Description: Patients with predominant amyloid kidney involvement at enrollment.
Time Frame: Data were assessed at baseline, 6 and 12 months, with change at end of study reported
Population: Analysis is limited to the patients with predominant amyloid kidney involvement at enrollment. Mixed models analyses of change from baseline levels of creatinine clearance (ml/min) and proteinuria (g/day) were performed to include all data collected at baseline, 6 and 12 months.
Measure: Mean (Standard Deviation); unit: g/day
Groups:
- Amyloid Nephropathy: Proteinuria (g/Day): Patients with predominant amyloid kidney involvement at enrollment.
Arm/Group | Amyloid Nephropathy: Proteinuria (g/Day)
Number analyzed (Participants) | 10
g/day | 5.91 (3.85)
Statistical Analysis 1: Comparison: Amyloid Nephropathy: Proteinuria (g/Day); Proteinuria (g/24 hours), baseline versus end study levels; Test type: Other — P-values and confidence intervals are not adjusted for multiple testing; p = 0.603, Mixed Models Analysis; degrees of freedom = 10; Change in outcome measure = 0.091, 95% CI 2-sided [-0.285 to 0.466]

ADVERSE EVENTS:
Groups:
- Doxycycline 100 mg po Bid x 12 Months: Open-label doxycycline 100 mg twice daily by mouth was administered to subjects for 12 months, if tolerated.
Arm/Group | Doxycycline 100 mg po Bid x 12 Months
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline 100 mg po Bid x 12 Months (N=25)
Fluid overload (Cardiac disorders) | 3 (4) — SOB, edema
Sun hypersensitivity (Skin and subcutaneous tissue disorders) | 1 (1) — Burns/desquamation induced by sun hypersensitivity
Bloating (Gastrointestinal disorders) | 1 (1) — Abdominal distension
Urinary retention (Renal and urinary disorders) | 1 (1)
osteonecrosis (Blood and lymphatic system disorders) | 1 (1)
Orthopedic issues (Surgical and medical procedures) | 2 (2)
Deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) — Ventricular trachycardia
Hip disease (Musculoskeletal and connective tissue disorders) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Skin cancer (Skin and subcutaneous tissue disorders) | 1 (1)
Hernia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline 100 mg po Bid x 12 Months (N=25)
Skin disruption (Skin and subcutaneous tissue disorders) | 15 (21)
GI disorder (Gastrointestinal disorders) | 9 (18)
Infection (Infections and infestations) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No